CLINICAL TRIAL: NCT07259811
Title: Vertebral Augmentation Using VCFix Spinal System in Stand-alone Configuration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amber Implants B.V. (Industry)
Collaborators: Avania B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-VS01-EU
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Vertebral Compression Fracture
Keywords: VCF; FIH; vertebral stabilization; fracture; trauma; osteoporosis; expandable implant
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VCFix Spinal System (Experimental)
  Interventions: Device: VCFix Spinal System in stand-alone configuration

INTERVENTIONS:
Device: VCFix Spinal System in stand-alone configuration — The distinguishing features of this intervention reside in: 1. In situ adjustment and maintenance of the height and angle of the device that allows expansion of the fractured VB in the cranio-caudal direction to realign the vertebral endplates and correct kyphosis. 2. The complex titanium perforated structure with optimized surface roughness that allows possible bone attachment, thereby permitting natural healing of the bone and potentially providing more stability to the device and the treated vertebra over time. 3. The ability to likely secure and reinforce the vertebra without using PMMA bone cement, avoiding all the symptomatic and asymptomatic side effects of bone cement. 4. The ability to connect the posterior to the anterior column of the spine through the pedicle screw component of the VCFix implant, therefore improving the biomechanical load distribution and consequently the ability to stabilize more severe fractures.

SUMMARY:
This study will review the safety and possibility of the VCFix Spinal System. This is a proof-of-concept study and an initial review of the surgical procedure and how well the VCFix device works, to who that the VCFix is safe and works well in early testings, so that a larger safety study can be done later to help get CE approval. The VCFix Spinal System will be used in its independent setup, within its planned use for treatment of vertebral compression fracture. It's designed to be a small early study to test safety and see if the treatment idea is possible, with one group and no blinding. Two hospitals in EU will enroll in total 10 participants with a single vertebral fracture that will undergo the same surgery.

The main test goals are: how successful the access creation of the vertebral body is using the VCFix Preparation kit according to the provided instructions, how successful the positioning of the VCFix implant is by using the VCFix Implantation kit according to the provided instructions, and how successful the fracture reduction by expanding the VCFix implant according to the provided instructions. The main safety goal is: number of device-/procedure-related major side effects through 30 days after the initial procedure.

Participant enrollment will last around 12 months. Each participant will be followed for 2 years after the implantations. All side effects related to the spine will be documented throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between 22 and 85 years of age
* One (single) vertebral fracture which meets all the following criteria:

  * Type A fractures as defined by the AO spine classification (compression injuries)1
  * Vertebral fracture located in the thoracic and lumbar regions of the spine
  * Fracture age <6 weeks or fractures with anatomic signs of reducibility (based on radiographic evidence as well as patient history)
  * Vertebral fracture shows an estimated height loss in the anterior or mid third of the vertebral body (VB) of at least 10% but not more than 70% based on radiographic evidence
  * Target VB has appropriate anatomy, i.e., suitable pedicle diameter, pedicle length and chord length that would allow for selection of correct implant size, as described in the IFU and based on axial MRI/CT scan before surgery Patient has a Numerical Pain Rating Scale (NPRS) back pain score of ≥5
* Patient has an Oswestry Disability Index (ODI) score of ≥30/100
* Patient has a BMI <35
* Patient is mentally capable of complying with trial protocol requirements for the duration of the study
* Patient can understand the risks and benefits of participating in the study and can provide written informed consent
* Patient is available for all study visits

Exclusion Criteria:

* Neoplasms with posterior involvement and/or presence of a mass within the spinal canal
* Non-mobile fractures (i.e., fracture is not recent (>6 weeks), bone marrow oedema or fluid or empty cleft are not visible in radiographic imaging, or fracture mode does not allow for fracture reduction in craniocaudal direction) 2
* Vertebral fracture prior to the incident fracture
* Fracture to the pedicle based on radiographic evaluation
* Asymptomatic vertebral fractures
* Patient clearly improving with pharmacological treatment
* Previous spine surgery, balloon kyphoplasty or vertebroplasty, for any vertebral fracture
* Spinal cord compression or canal compromise requiring decompression
* Severe back pain due to causes other than acute fracture with NPRS score > 5
* Pain due to any other condition that requires daily narcotic medication
* Pre-existing neurological deficit, radiculopathy or myelopathy
* Significant clinical comorbidity that the enrolling physician considers may either contraindicate surgery or interfere with long-term data collection or follow-up
* Pre-existing conditions such as:

  * Allergy to any components of the device/instruments used during the procedure or to PMMA bone cement
  * Active or incompletely treated infection of the vertebral column or active systemic infection, including unresolved urinary tract infection
  * Irreversible coagulopathy or bleeding disorder
  * Uncontrolled diabetes (HbA1c >8%)
  * Severe cardiopulmonary deficiencies
* Contraindications to MRI or radionuclide bone scan
* Concurrent participation in any other clinical study for which the primary outcomes are not achieved
* A life expectancy less than the study duration or undergoing palliative care
* Patient non-ambulatory prior to fracture
* Spondylolisthesis >Grade 1 at target vertebral body(s)
* Local kyphotic angle >30°
* Any underlying systemic bone disease other than osteoporosis (e.g., osteomalacia, osteogenesis imperfect, Paget's disease, etc.)
* The patient has pain based on clinical diagnosis of herniated nucleus pulposus or severe spinal stenosis (progressive weakness or paralysis)
* Any evidence of substance use disorder (alcohol, drugs)
* Ongoing long-term steroid therapy (steroid dose ≥30 mg /day for > 3 months)
* The patient is currently on anti-cancer therapy or anti-HIV therapy
* Patient known to be involved in medical litigation including Workmen's Compensation prior to the surgery
* Pregnancy or patients with child-bearing potential who do not accept taking contraception throughout the study duration
* Patients who require anterior stabilisation

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Outcome measure | 2 years
  Rate of successful vertebral body access creation through use of the VCFix Preparation kit according to the provided labelling
Outcome measure | 2 years
  Rate of successful positioning of the VCFix implant through use of the VCFix Implantation kit according to the provided labelling
Outcome measure | 2 years
  Rate of successful fracture reduction by expansion of the VCFix implant according to the provided labelling
Outcome measure | 30 days after index procedure
  Number of device-/procedure-related serious adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Wilhelmsburger Krankenhaus Groβ-Sand, Hamburg
  - Krankenhaus Mechernich, Mechernich

IPD SHARING:
Plan to Share IPD: No